CLINICAL TRIAL: NCT04908176
Title: A Drug-drug Interaction Study to Investigate the Effect of Avapritinib on the Pharmacokinetics of Midazolam in Patients With Unresectable or Metastatic Gastrointestinal Stromal Tumors (GIST) and Other Advanced Solid Tumors
Brief Title: A Drug-drug Interaction Study of Avapritinib and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BLU-285-1107
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Stromal Tumors; GIST; Non-resectable Advanced Solid Tumors; Recurrent or Unresectable Central Nervous System (CNS) Tumors
Keywords: Avapritinib; Midazolam; GIST; BLU-285; KIT; IDH-mutant astrocytoma; IDH-mutant oligodendroglioma; glioblastoma; H3K27-altered diffuse midline glioma; H3G34-mutant diffuse hemispheric glioma; midline glioma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Recurrence; Neoplasms; Glioblastoma | interventions — avapritinib; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with metastatic, unresectable GIST, non-CNS solid tumors, or CNS tumors (Experimental): Participants will receive 5 mg of midazolam orally on Day 1 and Day 17. Participants will receive avapritinib 300 mg daily, orally on starting on Day 3. Participants with CNS tumors will receive avapritinib 300 mg daily orally, until Day 56.
  Interventions: Drug: Avapritinib; Drug: midazolam

INTERVENTIONS:
Drug: Avapritinib — avapritinib tablets
  Other Names: BLU-285
Drug: midazolam — midazolam syrup

SUMMARY:
The purpose of this study is to investigate the effect of multiple dosing of avapritinib on the pharmacokinetics (PK) of midazolam in adult patients with metastatic or unresectable gastrointestinal stromal tumors (GIST), recurrent gliomas, or other KIT mutant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age at the time of signing the informed consent
2. Confirmed diagnosis of

   * metastatic or unresectable KIT mutant GIST that has recurred or progressed after at least 4 lines of prior systemic SOC therapy or the Investigator has determined that treatment with SOC therapy is not appropriate for patients who failed at least 2 lines of prior SOC

   OR

   ---Non-resectable advance solid tumor with KIT mutation with progression following standard of care treatment.

   OR

   ---Confirmed diagnosis of recurrent or unresectable CNS tumors including :IDH-mutant astrocytoma, IDH-mutant oligodendroglioma, glioblastoma, H3K27-altered diffuse midline glioma, H3G34-mutant diffuse hemispheric glioma, midline glioma (with unknown H3K27 mutation status) that has failed prior radiation or systemic SOC therapy.
3. Must be able to swallow an oral medication
4. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
5. Patient agrees to use contraception consistent with local regulations
6. Must provide signed informed consent to participate in the study

Exclusion Criteria:

1. Patients with GIST that harbors a known PDGFRA mutation
2. Known hypersensitivity to avapritinib, midazolam, or any of their excipients
3. Have received previous therapy with avapritinib
4. Have any of the following laboratory abnormalities before the first dose of study drug:

   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >3 × upper limit of normal (ULN) if no hepatic metastases are present; >5 × ULN if hepatic metastases are present
   * Total bilirubin >1.5 × ULN; >3 × ULN in the presence of Gilbert's Disease
   * Estimated (Cockcroft-Gault formula) or measured creatinine clearance <60 mL/min
   * Platelet count <100 × 10^9/liter (L)
   * Absolute neutrophil count (ANC) <1.0 × 10^9/L
   * Hemoglobin <9 grams per deciliter (g/dL). Transfusion and erythropoietin may be used to reach at least 9 g/dL but must have been administered at least 2 weeks before the first dose of the study drug.
5. Require therapy with a concomitant medication that is a strong and moderate CYP3A4 inhibitors or inducers
6. Consumption of any nutrients known to modulate CYP3A4 enzymes activity (eg, grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange and derivative products, cruciferous vegetables [eg, broccoli, cauliflower, cabbage, brussel sprouts]) within 14 days before screening and during the study until the end of the Main Treatment Period
7. Have received a prior anticancer drug less than 5 half-lives or 14 days (whichever is shorter) before screening
8. Have had a major surgical procedure within 14 days of the first dose of study drug or have significant traumatic injury within 28 days before screening
9. Have history of a cerebrovascular accident or transient ischemic attacks within 1 year before screening
10. Have known risk of intracranial bleeding, such as a brain aneurysm or history of subdural or subarachnoid bleeding
11. Have corrected QT interval using Fridericia's formula (QTcF) >450 msec
12. Have clinically significant, uncontrolled, cardiovascular disease, including congestive heart failure Grades 2, 3, or 4 according to the New York Heart Association classification, myocardial infarction, or unstable angina within the previous 6 months, or uncontrolled hypertension
13. Have experienced any hemorrhage or bleeding event National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 Grade ≥3 within 4 weeks before screening. Exceptions are patients with primary CNS tumors who are eligible if the Grade ≥3 bleeding event was in the CNS and it occurred 2 weeks or more prior to the first dose of avapritinib.
14. Patients who have a symptomatic nonhealing wound, ulcer, GI perforation, or bone fracture
15. Have received organ or allogenic bone marrow or peripheral blood stem cell transplant
16. Have known diagnosis of human immunodeficiency virus infection or active viral hepatitis; viral testing is not required
17. History of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink = 14 grams of alcohol). Alcohol consumption will be prohibited 48 hours before screening and throughout the entire the Main Treatment Period
18. Use of tobacco- or nicotine-containing products within 3 months of enrollment
19. Is a female patient who is unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for until at least 6 weeks after the last dose of study drug. Males who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of informed consent and for at least 6 weeks after the last dose of study drug.
20. Is a female patient who is pregnant, as documented by a serum beta human chorionic gonadotropin (β-hCG) pregnancy test consistent with pregnancy obtained within 7 days before the first dose of study drug. Patients with β-hCG values that are within the range for pregnancy but are not pregnant (false positives) may be enrolled with written consent of the Sponsor after pregnancy has been ruled out. Females of nonchildbearing potential (postmenopausal for more than 12 months, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) do not require a serum β-hCG test.
21. Female who is breastfeeding
22. Have a prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's opinion, could affect the safety of the patient, alter the absorption, distribution, metabolism or excretion of the study drugs, or impair the assessment of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration (Cmax) of midazolam | Day 1 and Day 18
time of maximum plasma concentration (tmax) of midazolam | Day 1 and Day 18
area under the plasma concentration-time curve (AUC) of midazolam | Day 1 and Day 18

SECONDARY OUTCOMES:
Number of adverse events (AEs), serious AEs (SAEs), | up to approximately 2 months
Cmax at steady state (Cmax, ss) of avapritinib | Day 18
Cmax at steady state (Cmax, ss) of metabolite | Day 18
area under the plasma concentration-time curve at steady state (AUC,ss) of avapritinib | Day 18
area under the plasma concentration-time curve at steady state (AUC,ss) of metabolite | Day 18

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No